CLINICAL TRIAL: NCT05188248
Title: A Pilot Study of the Immediate Effects of DLPFC tDCS on Attention Bias in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-01461
Record Dates: First submitted 2021-12-17; First posted 2022-01-12 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Female participants with Depression (Experimental): Female participants with mild to moderate depression to determine if a single-session of tDCS can alter negative attention bias. The primary objective is to study if single-session tDCS will affect attention bias in depression and is not meant to treat depression.
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Participants will complete a single 30 minutes tDCS session targeting the left DLPFC while sitting in a comfortable position. At the end of the tDCS session possible side effects experienced during the tDCS session will be recorded along with their intensity (rated using the visual analogue scale, 0-10) and duration. The session can be aborted at any time for any reason if the participant wishes.The MINDD STIM tDCS system is composed of a management component, treatment module, single-use sponge patches and supporting patches, a headband to hold in position the sponge patches, and 2 cables. A trained study technician will program the stimulation device through the management component setting to the following stimulation parameters:Stimulation intensity: 2.0 mA or 1.5 mA; Stimulation duration: 30 minutes;Ramp up duration: 30 seconds (beginning of stimulation);Ramp down duration: 30 seconds (end of stimulation)

SUMMARY:
Depression and other psychiatric conditions are marked by exaggerated, preferential processing (or attention bias) of negative information relative to neutral or positive information. This depression-related attention bias can be measured using the Dot Probe task and Visual Search, that allow assessment of the degree to which one shows bias toward negative information in the presence of neutral or positive information. A clinically effective treatment for depression is noninvasive brain stimulation with transcranial direct current stimulation (tDCS), targeting the dorsolateral prefrontal cortex (DLPFC), delivered in repeated sessions across a period of time. The study will test the effect of a single session of DLPFC tDCS on attention bias in patients with mild to moderate depression.

DETAILED DESCRIPTION:
This prospective pilot study will recruit 25 female participants, ages 18-45 (inclusive), with mild to moderate depression (based on BDI-II score range 14-19 for mild and 20-28 for moderate) to determine if a single-session of tDCS can alter negative attention bias. The primary objective is to study if single-session tDCS will affect attention bias in depression and is not meant to treat depression. Subjects may or may not be receiving treatment for mild-moderate depression.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45
* Female
* Mild to moderate depression (determined by BDI-II scores of 14-19 and 20-28, respectively)
* If taking antidepressants, medication must be stable ≥ 30 days prior to screening

Exclusion Criteria:

* Wide-Range Achievement Test-Fourth Edition (WRAT-4) Reading Subtest standard score <85 (to ensure understanding of test procedures)
* Insufficient visual and motor ability to operate the intervention and assessments as judged by treating neurologist or study staff
* Primary psychiatric disorder other than depression (based on MINI)
* Primary neurologic condition that would prevent ability to participate (as determined by study clinician).
* History of head trauma in the last year
* Medical device implants in the head or neck
* History or current uncontrolled seizure disorder
* Current substance abuse disorder
* . Pregnant or lactating women
* Skin disorder/sensitive skin near stimulation locations

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to leigh.charvet@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Pilloni G, Cho H, Tian TE, Beringer J, Bikson M, Charvet L. Immediate and Differential Response to Emotional Stimuli Associated With Transcranial Direct Current Stimulation for Depression: A Visual-Search Task Pilot Study. Neuromodulation. 2024 Jun;27(4):759-765. doi: 10.1016/j.neurom.2023.07.006. Epub 2023 Aug 20. PMID 37598327

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Female Participants With Depression
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Female Participants With Depression
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory (BDI-II) Score
Description: Measured by the Beck Depression Inventory (BDI-II) which is a brief, criteria-referenced assessment for measuring depression severity. The BDI-II consists of 21 items to assess the intensity of depression. Each item is a list of four statements arranged in increasing severity about a particular symptom of depression. The items are scored as 0, 1, 2, or 3. The score range is 0-63. Conventional cutoffs are 0-9 for normal range, 10-18 for mild to moderate depression, 19-29 for moderate to severe depression, and 30-63 for severe depression.
Time Frame: Study tDCS Administration Visit (Day1), Pre-tDCS Administration Time (1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Female Participants With Depression
Number analyzed (Participants) | 21
score on a scale | 21.29 (5.29)

2. Primary Outcome: Analog Mood Scale (AMS) Anxiety Score
Description: Analog Mood Scale (AMS) Anxiety is a brief measure of positive and negative mood asking "How anxious are you?". Participants were told to indicate their present mood by identifying a location on a horizontal line divided into 30 equally distanced segments labeled 1 (not at all) to 30 (very much). Higher scores indicated greater level of anxiety.
Time Frame: Study tDCS Administration Visit (Day1), Pre-tDCS Administration Time (1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Female Participants With Depression
Number analyzed (Participants) | 21
score on a scale | 7.95 (5.75)

3. Primary Outcome: Analog Mood Scale (AMS) Sad Score
Description: Analog Mood Scale (AMS) Sad is a brief measure of positive and negative mood asking "How sad are you?". Participants were told to indicate their present mood by identifying a location on a horizontal line divided into 30 equally distanced segments labeled 1 (not at all) to 30 (very much). Higher scores indicated greater level of sadness.
Time Frame: Study tDCS Administration Visit (Day1), Pre-tDCS Administration Time (1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Female Participants With Depression
Number analyzed (Participants) | 21
score on a scale | 7.19 (5.1)

4. Primary Outcome: Analog Mood Scale (AMS) Happy Score
Description: Analog Mood Scale (AMS) Happy is a brief measure of positive and negative mood asking "How happy are you?". Participants were told to indicate their present mood by identifying a location on a horizontal line divided into 30 equally distanced segments labeled 1 (not at all) to 30 (very much). Higher scores indicated greater level of happiness.
Time Frame: Study tDCS Administration Visit (Day1), Pre-tDCS Administration Time (1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Female Participants With Depression
Number analyzed (Participants) | 21
score on a scale | 11.67 (6.16)

5. Primary Outcome: Change in Analog Mood Scale (AMS) Anxiety Score
Description: Analog Mood Scale (AMS) Anxiety is a brief measure of positive and negative mood asking "How anxious are you?". Participants were told to indicate their present mood by identifying a location on a horizontal line divided into 30 equally distanced segments labeled 1 (not at all) to 30 (very much). Higher scores indicated greater level of anxiety. The AMS Anxiety will be administered before and after the Transcranial direct current stimulation (tDCS) session. The change in AMS Anxiety scores (Pre-tDCS Administration Time (1 hour) minus Post-tDCS Administration Time (1 hour)) is reported. A positive value indicates an improvement, less anxiety post-tDCS administration. A negative value indicates increased anxiety post-tDCS administration.
Time Frame: Pre-tDCS Administration Time (1 hour) and Post-tDCS Administration Time (1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Female Participants With Depression
Number analyzed (Participants) | 21
score on a scale | 2.76 (2.8)

6. Primary Outcome: Change in Analog Mood Scale (AMS) Sad Score
Description: Analog Mood Scale (AMS) Sad is a brief measure of positive and negative mood asking "How sad are you?". Participants were told to indicate their present mood by identifying a location on a horizontal line divided into 30 equally distanced segments labeled 1 (not at all) to 30 (very much). Higher scores indicated greater level of sadness. The AMS Sad will be administered before and after the Transcranial direct current stimulation (tDCS) session. The change in AMS Sad scores (Pre-tDCS Administration Time (1 hour) minus Post-tDCS Administration Time (1 hour)) is reported. A positive value indicates an improvement, less sadness post-tDCS administration. A negative value indicates increased sadness post-tDCS administration.
Time Frame: Pre-tDCS Administration Time (1 hour) and Post-tDCS Administration Time (1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Female Participants With Depression
Number analyzed (Participants) | 21
score on a scale | 2.62 (2.7)

7. Primary Outcome: Change in Normalized Response Time
Description: The Visual Search task will be administered to further assess attention bias, particularly examining the interference and facilitation effects in attention using emotional stimuli. The task uses emotional faces or words as stimuli, where the participant is instructed to search for the face that does not fit into the search set with respect to gender, where the target and distractors are expressing different or same emotions. This study will use this task as an outcome measure of Attention Bias. For this task, the change in mean response time (the time between display onset and button press) to the target stimulus is measured as the main outcome variable.
Time Frame: Pre-tDCS Administration Time (1 hour) and Post-tDCS Administration Time (1 hour)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Female Participants With Depression
Number analyzed (Participants) | 21
milliseconds | -0.39 (0.6)

ADVERSE EVENTS:
Time Frame: Right after the end of the 30-minute tDCS session
Arm/Group | Female Participants With Depression
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT05188248/Prot_SAP_000.pdf